CLINICAL TRIAL: NCT01428739
Title: Correlation Between MRS (Magnetic Resonance Spectroscopy) and Tumor Response to Radiation Therapy in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23701
Record Dates: First submitted 2010-10-21; First posted 2011-09-05 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2014-10

CONDITIONS: Breast Cancer
Keywords: cancer; MRS; Treatment response
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: MRS — Procedure
  Other Names: Philips 3 Tesla MRI Scanner

SUMMARY:
Correlation between MRS and Tumor Response Therapy in Breast Cancer.

DETAILED DESCRIPTION:
Correlation between MRS (Magnetic Resonance Spectroscopy and Tumor Response to Radiation in Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosed Breast cancer
* Patient is 18 years or older
* Karnofsky performance score > 70
* No previously irradiated or recurrent breast cancer
* No contraindication to MRS/MRI
* Signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
MRS Correlation with Treatment Response | Up to One Year
  measuring choline, water and fat levels by proton magnetic resonance spectroscopy in breast tumors in response to treatment

SECONDARY OUTCOMES:
Correlation with Tumor Stage | Up to One year

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Pervez, MBBS, FFRRCSI, FRCPC, Principal Investigator — Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada